CLINICAL TRIAL: NCT03996330
Title: The Taqman Microarray Card for Rapid Pathogen Identification in Ventilated Patients With Pneumonia
Brief Title: Rapid Pathogen Identification in Ventilated Patients With Pneumonia
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); Public Health England (Other Government)
Responsible Party: Principal Investigator, Andrew Conway Morris, Senior Research Associate and Honorary Consultant, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: 228951
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Pneumonia; Mechanical Ventilation Complication
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — broncho-alveolar lavage, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: taqman array card — The array card contains multiple PCR reactions for microbial pathogens, extracted microbial nuclear material from lavage or blood is run on the card to detect pathogen specific sequences by polymerase chain reaction.

SUMMARY:
Pneumonia, a serious infection of the lungs, is a common reason for Intensive Care Unit (ICU) admission. It may also develop as a significant complication of being on a mechanical ventilator. Although the clinical diagnosis is generally straight-forward to make, determining which organism is causing the infection (pathogen) presents a much greater challenge. Existing detection of pathogens relies on growing the organism under specific conditions in a microbiology laboratory. This process is slow, typically taking 48 to 72 hours, and is influenced by factors such as presence of antibiotics and the ease with which specific organisms can be grown. Conventional microbiology may only be positive less than 40% of cases of pneumonia and this means that patients are often treated with 'best guess' antibiotics. These antibiotics are generally broad spectrum, and risk the development of antibiotic resistance. Equally, organisms which are less commonly seen may not be covered by the initial antibiotic selection and may only be started once this organism is grown after 48 to 72 hours leading to delays in appropriate treatment. The aim of this study is to evaluate the performance of a new form of diagnostic test, using detection of pathogens by gene analysis rather than relying on growth. The investigators believe that this approach will be more rapid and more sensitive, and therefore likely to translate into more rapid and appropriate use of antibiotics.

DETAILED DESCRIPTION:
Pneumonia is a common cause of admission to the intensive care unit, and can also develop as a secondary complication of mechanical ventilation. The diagnosis of pneumonia relies on a combination of clinical and radiographic signs, demonstrating an inflammatory infiltrate to the lung parenchyma combined with evidence of infection. The treatment is appropriate antibiotics, together with supportive care as required by the patient's condition.

The selection of appropriate antibiotics presents a significant challenge, as between 60 and 70% of cases of pneumonia do not yield positive results on microbial cultures. This is the case in both community acquired and hospital acquired pneumonia. It can take up to 72 hours for results of conventional cultures to be returned, and these two aspects mean that pneumonia is commonly treated with empiric broad spectrum antibiotics. Rapid, sensitive tests for microbes could lead to a significant reduction in antibiotic use 1 and use of narrower spectrum agents, which will reduce the selective pressure for anti-microbial resistant organisms.

The investigators on this study have previously shown that a multiplex polymerase chain reactions targeting respiratory pathogens can enhance the detection of such organisms in patients with community-acquired pneumonia and immuno-compromised patients developing pneumonia. The use of a TaqMan microarray card allows for large multiplexing of the PCR reactions, which would allow a single card to target a wide range of potential respiratory pathogens including both community-acquired and hospital-acquired organisms.

The aim of this study is to evaluate a new taqMan multiplex PCR array card, which targets common community and hospital-acquired respiratory pathogens. The investigators anticipate that the results from this card will be available more rapidly than conventional culture. The investigators also aim to evaluate the diagnostic performance of the card, compared to conventional cultures, and validate its use in the population of ventilated patients in intensive care. In addition, conventional cultures of blood have a significantly lower yield in pneumonia that respiratory samples, however as they are considerably less invasive to obtain than broncho-alveolar lavage it would be advantageous if a highly sensitive assay for bacteria could detect relevant respiratory pathogen DNA in the blood. Therefore alongside the testing of respiratory samples, the investigators will assess the ability of the taqMan array to detect organisms in a contemporaneously obtained blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Mechanically ventilated
* Treating clinician clinically suspects pneumonia and is planning to undertake diagnostic bronchoscopy and lavage

Exclusion Criteria:

• Inability to gain advice from a personal or professional consultee. Where a patient has capacity, declining consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients in intensive care with suspected pneumonia, from community acquired, hospital acquired and ventilator-associated sources.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Time to result relative to conventional microbial culture | 5 days
  Comparison of the time to result returned to clinicians between the taqman array card and conventional microbial culture
Diagnostic performance compared to conventional culture | 5 days
  Comparison of sensitivity and negative predictive value of array card relative to conventional microbial culture

SECONDARY OUTCOMES:
Number and nature of organisms detected on taq-man array and not detected by conventional culture | 5 days
  Description of organisms detected on taq-man array and not detected by conventional culture
Sensitivity of PCR from blood relative to bronchoalveolar lavage PCR | 24 hours
  Comparison of the results of detection from broncho-alveolar lavage and blood

CONTACTS AND LOCATIONS:
Overall Officials: Vilas Navapurkar, MB ChB, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambs, United Kingdom

IPD SHARING:
Plan to Share IPD: No